CLINICAL TRIAL: NCT05557474
Title: Development and Clinical Validation of Early-stage Lung Cancer Prognostic Kit and Immunotherapy Companion Diagnostic Laboratory Developed Tests
Brief Title: Development and Clinical Validation of Early-stage Lung Cancer Prognostic Kit
Status: Recruiting | Type: Observational
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gee-Chen Chang, Chung Shan Medical University, Chung Shan Medical University
Other Study IDs: 110WFD2510303
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Surgery; Recurrence
Keywords: Lung Cancer; Immunohistochemistry; Enzyme-linked Immunosorbent Assay; Laboratory developed tests; Recurrence
MeSH Terms: conditions — Lung Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung cancer post surgery recurrence follow up: Lung adenocarcinoma, stage IA/IB/II/IIIA post-surgery follow up
  Interventions: Other: Early-stage lung cancer prognostic kit -- ELISA; Other: Early-stage lung cancer prognostic kit -- IHC

INTERVENTIONS:
Other: Early-stage lung cancer prognostic kit -- ELISA — blood sample with ELISA
Other: Early-stage lung cancer prognostic kit -- IHC — surgical tumor part with IHC

SUMMARY:
Lung cancer is the leading cause of cancer mortality worldwide in spite of the advanced progresses in medication and low-dose CT screening. The early-stage lung cancer accounts for less than 50% of newly diagnosed lung cancer in Taiwan, even in stage IB patients proximately 30% still suffer from recurrence and metastasis.

The International Cancer Moonshot Project recently established the first comprehensive proteogenomics profiling of early-stage lung cancer patients in East Asia, revealing a proteomics-informed classification to identify a new "late like" subtype, which can identify a subgroup of early-stage patients with worse clinicopathological features (Cell, Cover story, 2020). This study has been featured in prestigious journals (Nat Rev Clin Oncol; Cancer Discov, 2020) and led to two provisional US patents. In this proposal, taking the discovery from the Cancer Moonshot multiomics database, the investigators aim to translate these findings into clinical utilities. Two subprojects are proposed. (1) Validation of "late-like" protein markers for identifying high-risk early-stage lung cancer: Two IVD kits will be developed, including high-risk early-stage lung cancer IHC prediction kit for tumor staining and high-risk early lung cancer ELISA prediction kit for noninvasive diagnosis. (2) Conducting a prospective clinical trial to evaluate the accuracy of high-risk early-stage lung cancer IHC prediction kit and high-risk early-stage lung cancer ELISA prediction kit.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign and provide subject consent.
* Male or female of age 20 or older.
* Patients diagnosed with lung adenocarcinoma by tumor pathology.
* Lung cancer with the pathological stage of IA/IB/II/IIIA according to the American Joint Committee on Cancer Staging Manual (8th Edition).
* Complete tumor resection (R0 resection).
* The East Coast Cancer Clinical Research Collaborative (ECOG) performance status was 0 or 1 at the time of grouping.
* Those willing to provide tumor tissue or cytology specimens (including surgical specimens, tissue biopsy specimens, or cytology specimens), blood and body fluid specimens (for follow-up or disease recurrence, such as urine, malignant pleural effusion, ascites, pericardial fluid, etc.).

Exclusion Criteria:

* Not primary lung cancer patients.
* Lung cancer patients whose pathological stage is not IA/IB/II/IIIA according to the American Joint Committee on Cancer Staging Manual (8th Edition) after surgery.
* Patients with uncontrolled malignant tumors other than lung cancer.
* Uncontrolled systemic disease (such as diabetes, hypertension, active infection, etc.) (determined by the principal investigator )
* Pregnant women.
* Any condition may put the patient at serious risk, may affect the interpretation of the trial results, or may seriously interfere with the patient's participation in the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage lung adenocarcinoma post-surgical follow up
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  Disease free survival

SECONDARY OUTCOMES:
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chung Shan Medical University Hospital, Taichung, Taiwan
  - National Taiwan University, Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galon J, Bruni D. Tumor Immunology and Tumor Evolution: Intertwined Histories. Immunity. 2020 Jan 14;52(1):55-81. doi: 10.1016/j.immuni.2019.12.018. PMID 31940273
- [Background] Yarchoan M, Johnson BA 3rd, Lutz ER, Laheru DA, Jaffee EM. Targeting neoantigens to augment antitumour immunity. Nat Rev Cancer. 2017 Apr;17(4):209-222. doi: 10.1038/nrc.2016.154. Epub 2017 Feb 24. PMID 28233802
- [Background] Chen YJ, Roumeliotis TI, Chang YH, Chen CT, Han CL, Lin MH, Chen HW, Chang GC, Chang YL, Wu CT, Lin MW, Hsieh MS, Wang YT, Chen YR, Jonassen I, Ghavidel FZ, Lin ZS, Lin KT, Chen CW, Sheu PY, Hung CT, Huang KC, Yang HC, Lin PY, Yen TC, Lin YW, Wang JH, Raghav L, Lin CY, Chen YS, Wu PS, Lai CT, Weng SH, Su KY, Chang WH, Tsai PY, Robles AI, Rodriguez H, Hsiao YJ, Chang WH, Sung TY, Chen JS, Yu SL, Choudhary JS, Chen HY, Yang PC, Chen YJ. Proteogenomics of Non-smoking Lung Cancer in East Asia Delineates Molecular Signatures of Pathogenesis and Progression. Cell. 2020 Jul 9;182(1):226-244.e17. doi: 10.1016/j.cell.2020.06.012. PMID 32649875
- [Background] Jamal-Hanjani M, Wilson GA, McGranahan N, Birkbak NJ, Watkins TBK, Veeriah S, Shafi S, Johnson DH, Mitter R, Rosenthal R, Salm M, Horswell S, Escudero M, Matthews N, Rowan A, Chambers T, Moore DA, Turajlic S, Xu H, Lee SM, Forster MD, Ahmad T, Hiley CT, Abbosh C, Falzon M, Borg E, Marafioti T, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Shah R, Joseph L, Quinn AM, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Dentro S, Taniere P, O'Sullivan B, Lowe HL, Hartley JA, Iles N, Bell H, Ngai Y, Shaw JA, Herrero J, Szallasi Z, Schwarz RF, Stewart A, Quezada SA, Le Quesne J, Van Loo P, Dive C, Hackshaw A, Swanton C; TRACERx Consortium. Tracking the Evolution of Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 1;376(22):2109-2121. doi: 10.1056/NEJMoa1616288. Epub 2017 Apr 26. PMID 28445112